CLINICAL TRIAL: NCT00000898
Title: A Prototype Study to Test the Effect of Staggered Dosing on the Pharmacokinetic Interactions Between Paired Combinations of Nelfinavir (NFV), Ritonavir (RTV), and Soft Gelatin Capsule of Saquinavir (SQVsgc)
Brief Title: The Effects of Staggered Dosing on Interactions Between Paired Combinations of Nelfinavir, Ritonavir, and Saquinavir
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 378; 11339 (Registry Identifier: DAIDS ES)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Drug Interactions; Drug Therapy, Combination; Saquinavir; HIV Protease Inhibitors; Ritonavir; Nelfinavir
MeSH Terms: conditions — HIV Infections | interventions — Ritonavir; Nelfinavir; Saquinavir

INTERVENTIONS:
Drug: Ritonavir
Drug: Nelfinavir mesylate
Drug: Saquinavir

SUMMARY:
The purpose of this study is to see if staggering doses of nelfinavir, ritonavir, and saquinavir has any effect on the interactions between these drugs.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Absence of HIV-1 infection as documented by any licensed ELISA test kit within 14 days prior to study entry.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms and conditions are excluded:

* Any medical condition that, in the opinion of the investigator, would interfere with the patient's ability to participate in this protocol.

Patients with the following prior conditions and symptoms are excluded:

* History of chronic illness such as hypertension, coronary artery disease, arthritis, diabetes, or any chronic gastrointestinal conditions that might interfere with drug absorption.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18
Dates: Study Completion 2000-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Blaschke T, Study Chair; Flexner C, Study Chair; Sheiner L, Study Chair
Locations (4):
- United States (4):
  - San Francisco Gen Hosp, San Francisco, California
  - Univ of California/ San Francisco / Dept of Medicine, San Francisco, California
  - Stanford Univ Med Ctr, Stanford, California
  - Johns Hopkins Hosp, Baltimore, Maryland

REFERENCES:
- [Background] Washington CB, Flexner C, Sheiner LB, Rosenkranz SL, Segal Y, Aberg JA, Blaschke TF; AIDS Clinical Trials Group Protocol (ACTG 378) Study Team. Effect of simultaneous versus staggered dosing on pharmacokinetic interactions of protease inhibitors. Clin Pharmacol Ther. 2003 May;73(5):406-16. doi: 10.1016/s0009-9236(03)00006-7. PMID 12732841